CLINICAL TRIAL: NCT00441805
Title: The Treatment of Acne Vulgaris With Radiofrequency Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated- the study was not started (per Investigator's/sponsor decision)
Sponsor: Alma Lasers (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-RF/ACN02/06IL CTIL
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Acne Vulgaris
Keywords: Acne; RadioFrequency
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Radio Frequency

SUMMARY:
Radiofrequency emmitting device, normaly used for thermage treatments will be used on 22 mild to moderate acne patients faces.

The aim of the study is to check whether RF heating of subcutaneous and dermis will improve acne in needed patients.

ELIGIBILITY:
Inclusion Criteria:

* mild-moderate Acne
* age over 18
* otherwise healthy

Exclusion Criteria:

* age under 18
* pregnancy
* systemic acne treatment in the last month
* local acne treatment in the last month

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-11 (Estimated); Primary Completion 2007-09 (Estimated); Study Completion 2007-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yussi Levcelter, Dr., Study Director — Alma Lasers LTD
Locations (1):
- Lase Ohr clinic, Jerusalem, Israel